CLINICAL TRIAL: NCT06222684
Title: The Effect of Music on Pain, Anxiety and Satisfaction During Mammography
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Sümeyye Köse, Phd Student, Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: SumeyyeKose
Record Dates: First submitted 2024-01-09; First posted 2024-01-25 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Breast Cancer; Pain; Anxiety
Keywords: mammography; pain; music therapy
MeSH Terms: conditions — Breast Neoplasms; Pain; Anxiety Disorders | interventions — Music Therapy

STUDY DESIGN:
Intervention Model Description: The study is a randomized controlled trial.
Who Masked: Participant
Masking Description: The evaluation was made by the participants in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Women in the intervention group applying for mammography screening will listen to music for 5 minutes before, during and after the procedure.
  Interventions: Other: Music therapy
- Control Group (No Intervention): Women in the control group applying for mammography screening will not receive any intervention other than routine mammography screening.

INTERVENTIONS:
Other: Music therapy — Women applying for mammography screening will receive music therapy for 5 minutes before the procedure, during the mammography scan and for 5 minutes after the procedure.
  Arms: Intervention Group

SUMMARY:
This study was planned to determine the effect of music listened to during mammography screening on pain, anxiety and satisfaction.

DETAILED DESCRIPTION:
The randomized controlled and experimental study will be conducted with 70 women who apply to the Cancer Early Diagnosis, Screening and Training Center for mammography screening. Women in the experimental group (n=35) will listen to music before, during and after mammography screening, and women in the control group (n=35) will undergo routine mammography screening. Information Form Containing Sociodemographic Information and Situational Anxiety Inventory will be used to collect data.

ELIGIBILITY:
Inclusion Criteria:

* Knowing how to read and write,
* Not having had a mammogram before,
* Being between the ages of 40-69,
* No hearing-related problems,
* Not having used analgesic or anesthetic medication within 24 hours before or during the procedure,
* Voluntarily participating in the study,

Exclusion Criteria:

- The woman has a cognitive and auditory problem

Ages: 40 Years to 69 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-04-20 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Anxiety | 20 minutes
  Data will be collected using the State Anxiety Inventory. The answer options collected in four classes on the State Anxiety Inventory scale are: (1) Not at all, (2) A little, (3) A lot and (4) Completely; The options on the trait anxiety scale are (1) Rarel, (2) Sometimes, (3) A lot of the time, and (4) Almost always. The higher the score obtained from the scales, the higher the person's anxiety is. The total score obtained from the scale varies between 20-80, and 20-39 indicates a mild anxiety level, 40-59 indicates a medium anxiety level, 60-79 indicates a high anxiety level, and 80 points indicates a panic anxiety level.
Pain Level | 20 minutes
  Data will be collected using the Visual Analogue Scale. Pain can be given a score between 0 and 10 on the scale.The higher the scale score, the greater the pain.

SECONDARY OUTCOMES:
Satisfaction Level | 20 minutes
  Data will be collected using the Visual Analog Scale. Satisfaction can be given a score between 0 and 10 on the scale. The higher the scale score, the higher the satisfaction level.

CONTACTS AND LOCATIONS:
Locations (1):
- Pendik District Health Directorate Maternal Child Health and Family Planning Center, Istanbul, Pendik, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No